CLINICAL TRIAL: NCT06860919
Title: Evaluation Prospective Des résultats du Suivi Pluridisciplinaire Mis en Place au décours d'Une Consultation de Transition Pour l'atrésie de l'œsophage
Brief Title: Prospective Evaluation of the Results of Multidisciplinary Follow-up After a Transitional Consultation for Esophageal Atresia
Acronym: TAO
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240714
Record Dates: First submitted 2025-01-16; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-01

CONDITIONS: Esophageal Atresia
Keywords: Esophageal Atresia
MeSH Terms: conditions — Esophageal Atresia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Young adults with esophageal atresia
  Interventions: Other: Follow-up of the patients during 3 years

INTERVENTIONS:
Other: Follow-up of the patients during 3 years — Evaluation of PTSD prevalence, anxiety-depressive state, quality of life, look for a correlation between their clinical history and PTSD.
  Analysis of the nutritional, gastrointestinal and respiratory status.

SUMMARY:
A transition consultation for adult patients with esophageal atresia, involving medical and paramedical stakeholders, was set up at Hôpital Saint-Louis in 2020. The aim of this initiative is to: 1. initiate adult medical, psychological and social follow-up; 2. empower these adults in their future care; 3. establish a personalized follow-up schedule. This project is the first to focus on post-traumatic stress disorder (PTSD) in young adults with esophageal atresia. A 3-year analysis of the somatic and psychosocial variables analyzed will confirm the validity of this initiative, and define its optimal contours for improving these patients' quality of life as adults.

ELIGIBILITY:
Inclusion Criteria:

* Patients with esophageal atresia
* Aged 18 to 30
* Followed at Hôpital Saint Louis
* Informed and not opposed to the study
* Patients affiliated to a social security scheme

Exclusion Criteria:

* Inability to answer questionnaires
* Patients under guardianship
* Patients under AME (Aide Médicale d'Etat in France)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young adults with esophageal atresia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2030-12-19 (Estimated); Study Completion 2030-12-19 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Post Traumatic Stress Disorder | At day 0

SECONDARY OUTCOMES:
Hospital Anxiety and Depression score | At day 0
  The HAD scale is a self-assessment scale for detecting states of depression and anxiety in the setting of an hospital medical outpatient clinic.
  HAD scale is a self-administered scale of 14 items which assessed levels of depression and anxiety, divided into 2 subscales of 7 items (Anxiety or HADS-A, Depression or HADS-D). Each item is scored on a scale of 0 to 3. A score is generated for each of the two sub-scales (sum of the 7 items, ranging from 0 to 21). A higher score indicates worse outcome.
Hospital Anxiety and Depression score | At 3 years
  The HAD scale is a self-assessment scale for detecting states of depression and anxiety in the setting of an hospital medical outpatient clinic.
  HAD scale is a self-administered scale of 14 items which assessed levels of depression and anxiety, divided into 2 subscales of 7 items (Anxiety or HADS-A, Depression or HADS-D). Each item is scored on a scale of 0 to 3. A score is generated for each of the two sub-scales (sum of the 7 items, ranging from 0 to 21). A higher score indicates worse outcome.
Quality of life evaluation | At day 0
  EA QOL questionnaire The score includes 4 domains : eating, social relationships, body perception, and health and well-being.
  The score varies between 0 to 100, the higher score the higher the quality of life.
Quality of life evaluation | At 3 years
  EA QOL questionnaire The score includes 4 domains : eating, social relationships, body perception, and health and well-being.
  The score varies between 0 to 100, the higher score the higher the quality of life.
Eating assessment | At day 0
  EAT-10 is an auto-questionnaireto evaluate dysphagia. There are 10 items, with a result for each varying between 0 (no problem) and 4 (severe problems)
Eating assessment | At 3 years
  EAT-10 is an auto-questionnaireto evaluate dysphagia. There are 10 items, with a result for each varying between 0 (no problem) and 4 (severe problems)
Quality of life assessment | At day 0
  It will be assessed by the SF36 scale. The Short Form (36) Health Survey is a 36-item measure if health status. The score obtained varies between 0 and 100. The higher the score the less disability.
  Ware JE, Sherbourne CD. The MOS 36-item short-form health survey (SF-36): I. Conceptual framework and item selection. Med Care 1992;30:473-83.
Quality of life assessment | At 3 years
  It will be assessed by the SF36 scale. The Short Form (36) Health Survey is a 36-item measure if health status. The score obtained varies between 0 and 100. The higher the score the less disability.
  Ware JE, Sherbourne CD. The MOS 36-item short-form health survey (SF-36): I. Conceptual framework and item selection. Med Care 1992;30:473-83.
Weight | At day 0
Weight | At 3 years
Height | At day 0
Height | At 3 years
Body Mass Index | At day 0
Body Mass Index | At 3 years
thoracic CT scan | At day 0
thoracic CT scan | At 3 years
respiratory function test | At day 0
respiratory function test | At 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Saint Louis, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided